CLINICAL TRIAL: NCT03376516
Title: Clinical Study to Investigate the Pharmacokinetics, Efficacy, Safety, and Immunogenicity of Wilate in Previously Treated Paediatric Patients With Severe Haemophilia A
Brief Title: Pharmacokinetics, Efficacy, Safety, and Immunogenicity of Wilate in Previously Treated Paediatric Patients With Severe Haemophilia A
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Octapharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WIL-30
Record Dates: First submitted 2017-12-13; First posted 2017-12-18 (Actual); Results first posted 2019-12-24 (Actual); Last update posted 2021-01-19 (Actual); Status verified 2020-12

CONDITIONS: Severe Hemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — von Willebrand Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- All patients (Experimental): All patients will receive Wilate for prophylactic treatment. Patients will also receive Wilate for treatment of breakthrough bleeding events as required
  Interventions: Drug: Wilate

INTERVENTIONS:
Drug: Wilate — von Willebrand factor / Factor VIII (plasma derived)

SUMMARY:
A prospective, non-controlled, international, multi-centre phase 3 study to investigate the pharmacokinetics, efficacy, safety, and immunogenicity of Wilate in previously treated children with severe haemophilia A

ELIGIBILITY:
Inclusion Criteria:

1. Severe haemophilia A (<1% FVIII:C) according to medical history
2. Male patients aged 1 to <12 years
3. Previous treatment with a FVIII concentrate for at least 50 exposure days (EDs)
4. Immunocompetence (CD4+ count >200/μL)
5. Voluntarily given, fully informed written and signed consent obtained by the patient's parent(s) or legal guardian and, depending on the children's developmental stage and intellectual capacity, informed assent by the patients before any study-related procedures are performed

The interval between the Screening Visit and the PK Visit should not exceed 30 days. If the 30-day interval is exceeded, determination of the CD4+ count is to be repeated and must be >200/μL for patients to be enrolled (i.e., inclusion criterion no. 4).

Exclusion Criteria:

1. Any coagulation disorders other than haemophilia A
2. History of FVIII inhibitor activity (≥0.6 BU) or detectable FVIII inhibitory antibodies (≥0.6 BU using the Nijmegen modification of the Bethesda assay) at screening, as determined by the central laboratory
3. Severe liver or kidney diseases (alanine aminotransferase [ALAT] and aspartate transaminase [ASAT] levels >5 times of upper limit of normal, creatinine >120 μmol/L)
4. Patients receiving or scheduled to receive immunomodulating drugs (other than antiretroviral chemotherapy), such as alpha-interferon, prednisone (equivalent to >10 mg/day), or similar drugs

Ages: 1 Year to 11 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 11 (Actual)
Dates: Start 2017-11-22 (Actual); Primary Completion 2018-11-03 (Actual); Study Completion 2018-11-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Solomon, MD, Study Director — Octapharma
Locations (3):
- Kirov SSC Hematology and Transfusiology, Kirov, Russia
- Ukraine (2):
  - "National Children's Specialized Clinic "OKHMATDYT", Kyiv
  - "Western Ukrainian Specialized Children's Medical Center", Lviv

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Wilate: A total of 11 patients were enrolled in this study. For the pharmacokinetic (PK) assessment a single dose of Wilate (50±5 IU/kg BW) was administered to 10 patients.
  Prophylactic treatment: Wilate (20-40 IU/kg BW) was administered every 2-3 days for 6 months. In case of unacceptably frequent spontaneous breakthrough bleeding episodes (BEs) the dose of Wilate was to be increased by approximately 5 IU/kg.
  The dose (and duration) of treatment for breakthrough BEs was dependent on the location and extent of bleeding and on the clinical condition of the patient; range: 10-50 IU/kg every 12-24 hours or 8-24 hours until resolved.
  Two patients underwent surgery treated with Wilate (SURG population). Minor surgeries received 15-30 IU/kg of Wilate every 24 hours until healing was achieved. Major surgeries were treated with 40-50 IU/kg, repeat injection every 8-24 hours until adequate wound healing, then therapy for at least another 7 days to maintain a FVIII activity of 30% to 60%.
Period: Overall Study
Arm/Group | Wilate
Started | 11
Received Treatment | 10
SAF Population (SAF population = study population of patients in safety analysis) | 10
FAS Population (FAS population = full analysis population) | 10
PK Population (PK population = study population of patients who underwent pharmacokinetic analysis) | 10
PP Population (PP population = per-protocol population) | 9
SURG Population (SURG population = study population of patients undergoing surgery treated with Wilate) | 2
Completed | 9
Not Completed | 2
Not completed — Not treated | 1
Not completed — Consent withdrawn | 1

BASELINE CHARACTERISTICS:
Population: The safety (SAF) population included all patients who received at least one injection of Wilate during the study (n=10).
Groups:
- Wilate: The safety (SAF) population includes all patients who received at least one injection of Wilate during the study (n=10).
Arm/Group | Wilate
Number analyzed (Participants) | 10
Age, Customized [Mean (Standard Deviation); unit: years] — Age at screening (years) Population: The overall safety (SAF) population included all patients who received at least one injection of Wilate during the study (n=10). Of these, 5 patients aged 1-<6 years were analyzed, and 5 patients aged 6-<12 years were analyzed.
  years
    1-<6 years: number analyzed (Participants) | 5
    1-<6 years | 4.0 (1.2)
    6-<12 years: number analyzed (Participants) | 5
    6-<12 years | 9.8 (0.8)
    Total | 6.9 (3.2)
Sex/Gender, Customized [Count of Participants; unit: Participants] — Population: The overall safety (SAF) population included all patients who received at least one injection of Wilate during the study (n=10). Of these, 5 patients 1-<6 years were analyzed, and 5 patients aged 6-<12 years were analyzed.
  Participants
    1-<6 years: number analyzed (Participants) | 5
    1-<6 years: Female | 0
    1-<6 years: Male | 5
    6-<12 years: number analyzed (Participants) | 5
    6-<12 years: Female | 0
    6-<12 years: Male | 5
    Total: Female | 0
    Total: Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: The overall safety (SAF) population included all patients who received at least one injection of Wilate during the study (n=10). Of these, 5 patients 1-<6 years were analyzed, and 5 patients aged 6-<12 years were analyzed.
  Participants
    1-<6 years: number analyzed (Participants) | 5
    1-<6 years: American Indian or Alaska Native | 0
    1-<6 years: Asian | 0
    1-<6 years: Native Hawaiian or Other Pacific Islander | 0
    1-<6 years: Black or African American | 0
    1-<6 years: White | 5
    1-<6 years: More than one race | 0
    1-<6 years: Unknown or Not Reported | 0
    6-<12 years: number analyzed (Participants) | 5
    6-<12 years: American Indian or Alaska Native | 0
    6-<12 years: Asian | 0
    6-<12 years: Native Hawaiian or Other Pacific Islander | 0
    6-<12 years: Black or African American | 0
    6-<12 years: White | 5
    6-<12 years: More than one race | 0
    6-<12 years: Unknown or Not Reported | 0
    Total: American Indian or Alaska Native | 0
    Total: Asian | 0
    Total: Native Hawaiian or Other Pacific Islander | 0
    Total: Black or African American | 0
    Total: White | 10
    Total: More than one race | 0
    Total: Unknown or Not Reported | 0
Weight [Mean (Standard Deviation); unit: kg] — Population: The overall safety (SAF) population included all patients who received at least one injection of Wilate during the study (n=10). Of these, 5 patients 1-<6 years were analyzed, and 5 patients aged 6-<12 years were analyzed.
  kg
    1-<6 years: number analyzed (Participants) | 5
    1-<6 years | 16.9 (3.6)
    6-<12 years: number analyzed (Participants) | 5
    6-<12 years | 37.4 (5.4)
    Total | 27.2 (11.6)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Population: The overall safety (SAF) population included all patients who received at least one injection of Wilate during the study (n=10). Of these, 5 patients 1-<6 years were analyzed, and 5 patients aged 6-<12 years were analyzed.
  kg/m^2
    1-<6 years: number analyzed (Participants) | 5
    1-<6 years | 15.3 (1.3)
    6-<12 years: number analyzed (Participants) | 5
    6-<12 years | 17.7 (2.2)
    Total | 16.5 (2.1)
Blood groups [Count of Participants; unit: Participants] — Population: The overall safety (SAF) population included all patients who received at least one injection of Wilate during the study (n=10). Of these, 5 patients 1-<6 years were analyzed, and 5 patients aged 6-<12 years were analyzed.
  Participants
    1-<6 years: number analyzed (Participants) | 5
    1-<6 years: O | 2
    1-<6 years: A | 1
    1-<6 years: AB | 0
    1-<6 years: B | 2
    6-<12 years: number analyzed (Participants) | 5
    6-<12 years: O | 2
    6-<12 years: A | 3
    6-<12 years: AB | 0
    6-<12 years: B | 0
    Total: O | 4
    Total: A | 4
    Total: AB | 0
    Total: B | 2
Previous Factor (F)VIII treatment [Count of Participants; unit: Participants] — Population: The overall safety (SAF) population included all patients who received at least one injection of Wilate during the study (n=10). Of these, 5 patients 1-<6 years were analyzed, and 5 patients aged 6-<12 years were analyzed.
  Participants
    1-<6 years: number analyzed (Participants) | 5
    1-<6 years: On-demand | 0
    1-<6 years: Prophylaxis | 3
    1-<6 years: Combination | 2
    6-<12 years: number analyzed (Participants) | 5
    6-<12 years: On-demand | 2
    6-<12 years: Prophylaxis | 0
    6-<12 years: Combination | 3
    Total: On-demand | 2
    Total: Prophylaxis | 3
    Total: Combination | 5
Previous annualised bleeding rate (ABR) [Mean (Standard Deviation); unit: Bleeding events per year (ABR)] — Previous ABR is based on the bleeding rate in the 6 months prior to entry into the study. Population: The overall safety (SAF) population included all patients who received at least one injection of Wilate during the study (n=10). Of these, 5 patients 1-<6 years were analyzed, and 5 patients aged 6-<12 years were analyzed.
  Bleeding events per year (ABR)
    1-<6 years: number analyzed (Participants) | 5
    1-<6 years | 4.8 (3.0)
    6-<12 years: number analyzed (Participants) | 5
    6-<12 years | 13.6 (8.9)
    Total | 9.2 (7.8)

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetic (PK) Assessment (Area Under the Curve (AUC)) of FVIII:C
Description: PK assessments of the factor VIII coagulant activity (FVIII:C) for Wilate were determined using the one-stage (OS) assay. The units of measure to calculate AUC is hours (h) x international units (IU)/decilitre (dL).
Time Frame: 0h, 0.25h, 1h, 6h, 24h and 48 h following a single dose of Wilate
Population: The analysis was performed in the PK population which included all patients who underwent PK assessment during the study (total: n=10). The PK population comprised 5 patients aged 1-<6 years and 5 patients aged 6-<12 years.
Measure: Mean (Standard Deviation); unit: h*IU/dL
Groups:
- Wilate: PK population
Arm/Group | Wilate
Number analyzed (Participants) | 10
h*IU/dL
  1-<6 years: number analyzed (Participants) | 5
  1-<6 years | 768.8 (288.5)
  6-<12 years: number analyzed (Participants) | 5
  6-<12 years | 671.9 (289.7)
  Total | 720.3 (277.3)

2. Primary Outcome: Pharmacokinetic (PK) Assessment (Area Under the Curve [AUC] Normalised (AUCNorm)) of FVIII:C for Wilate
Description: PK assessments of the factor VIII coagulant activity (FVIII:C) for Wilate were determined using the one-stage (OS) assay. The mean area under the curve normalised for the administered dose (AUCnorm) was calculated for Wilate.
  The units of measure used were AUC divided by dose.
Time Frame: 0h, 0.25h, 1h, 6h, 24h and 48 h following a single dose of Wilate
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h*kg/dL
Arm/Group | Wilate
Number analyzed (Participants) | 10
h*kg/dL
  1-<6 years: number analyzed (Participants) | 5
  1-<6 years | 15.38 (5.77)
  6-<12 years: number analyzed (Participants) | 5
  6-<12 years | 13.44 (5.79)
  Total | 14.41 (5.55)

3. Primary Outcome: Pharmacokinetic (PK) Assessment (Half-life (h)) of FVIII:C
Description: PK assessments of the factor VIII coagulant activity (FVIII:C) for Wilate were determined using the one-stage (OS) assay. The units of measure to calculate half-life is hours.
Time Frame: 0h, 0.25h, 1h, 6h, 24h and 48 h following a single dose of Wilate
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Wilate
Number analyzed (Participants) | 10
hours
  1-<6 years: number analyzed (Participants) | 5
  1-<6 years | 8.28 (1.51)
  6-<12 years: number analyzed (Participants) | 5
  6-<12 years | 9.35 (2.40)
  Total | 8.82 (1.97)

4. Primary Outcome: Pharmacokinetic (PK) Assessment (Maximum Plasma Concentration) for FVIII:C
Description: PK assessments of FVIII:C were determined using the one-stage (OS) assays. The maximum plasma concentration of FVIII:C was calculated based on the FVIII:C values measured in the patients participating in the PK study.
  Units of measure for maximum plasma concentration are international units (IU)/ decilitre (dL)
Time Frame: 0h, 0.25h, 1h, 6h, 24h and 48 h following a single dose of Wilate
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: IU/dL
Arm/Group | Wilate
Number analyzed (Participants) | 10
IU/dL
  1-<6 years: number analyzed (Participants) | 5
  1-<6 years | 83.0 (16.5)
  6-<12 years: number analyzed (Participants) | 5
  6-<12 years | 78.94 (26.56)
  Total | 80.99 (20.94)

5. Primary Outcome: Pharmacokinetic (PK) Assessment (Time to Reach Maximum Plasma Concentration (Tmax)) of FVIII:C
Description: PK assessments of the factor VIII coagulant activity (FVIII:C) for Wilate were determined using the one-stage (OS) assay. The units of measure to calculate Tmax is hours (h).
Time Frame: 48 h following a single dose of Wilate
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Wilate
Number analyzed (Participants) | 10
hours
  1-<6 years: number analyzed (Participants) | 5
  1-<6 years | 0.25 (0.00)
  6-<12 years: number analyzed (Participants) | 5
  6-<12 years | 0.25 (0.00)
  Total | 0.25 (0.00)

6. Primary Outcome: Pharmacokinetic (PK) Assessment (Mean Residence Time (MRT)) of FVIII:C
Description: PK assessments of the factor VIII coagulant activity (FVIII:C) for Wilate were determined using the one-stage (OS) assay. The units of measure to calculate MRT is hours.
Time Frame: 48 h following a single dose of Wilate
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Wilate
Number analyzed (Participants) | 10
hours
  1-<6 years: number analyzed (Participants) | 5
  1-<6 years | 11.47 (2.34)
  6-<12 years: number analyzed (Participants) | 5
  6-<12 years | 12.56 (3.53)
  Total | 12.01 (2.88)

7. Primary Outcome: Pharmacokinetic (PK) Assessment (Volume of Distribution (Vd)) of FVIII:C
Description: PK assessments of the factor VIII coagulant activity (FVIII:C) for Wilate were determined using the one-stage (OS) assay. The units of measure to calculate Vd is decilitre (dL)/ kilograms (kg).
Time Frame: 0h, 0.25h, 1h, 6h, 24h and 48 h following a single dose of Wilate
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: dL/kg
Arm/Group | Wilate
Number analyzed (Participants) | 10
dL/kg
  1-<6 years: number analyzed (Participants) | 5
  1-<6 years | 0.784 (0.177)
  6-<12 years: number analyzed (Participants) | 5
  6-<12 years | 1.081 (0.494)
  Total | 0.933 (0.384)

8. Primary Outcome: Pharmacokinetic (PK) Assessment (Clearance) of FVIII:C
Description: PK assessments of the factor VIII coagulant activity (FVIII:C) for Wilate were determined using the one-stage (OS) assay. The units of measure to calculate clearance are decilitre (dL)/ hours (h)/ kilograms (kg).
Time Frame: 0h, 0.25h, 1h, 6h, 24h and 48 h following a single dose of Wilate
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: dL/h/kg
Arm/Group | Wilate
Number analyzed (Participants) | 10
dL/h/kg
  1-<6 years: number analyzed (Participants) | 5
  1-<6 years | 0.071 (0.019)
  6-<12 years: number analyzed (Participants) | 5
  6-<12 years | 0.098 (0.074)
  Total | 0.084 (0.053)

9. Primary Outcome: Incremental In Vivo Recovery (IVR) of FVIII:C
Description: The incremental IVR was determined from all patients at baseline was determined using the one-stage (OS) assay (standardised to 50 IU/kg).
  The units of measure to calculate IVR is kilograms (kg) / deciliter (dL)
Time Frame: 48 h following a single dose of Wilate
Population: This analysis was performed for the full-analysis (FAS) population which included all patients who has at least one injection of Wilate (n=10). The FAS population comprised 5 patients aged 1-<6 years and 5 patients aged 6-<12 years.
Measure: Mean (Standard Deviation); unit: kg/dL
Groups:
- 1-<6 Years: FAS population patients aged 1-<6 years
- 6-<12 Years: FAS population patients aged 6-<12 years
- Total: All patients in the FAS population.
Arm/Group | 1-<6 Years | 6-<12 Years | Total
Number analyzed (Participants) | 5 | 5 | 10
kg/dL | 1.65 (0.33) | 1.57 (0.53) | 1.61 (0.42)

10. Secondary Outcome: Total Annualized Bleeding Rate (TABR)
Description: The total number of bleeding events (BEs) in the time period between the first dose of IMP and the study completion visit, divided by the duration (in years) between the first dose of IMP and the study completion visit.
  Surgery periods, and BEs occurring within these periods, will be excluded from the calculation of TABR.
Time Frame: 6 months
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Bleeding events per year (TABR)
Groups:
- Wilate: FAS population
Arm/Group | Wilate
Number analyzed (Participants) | 10
Bleeding events per year (TABR)
  1-<6 years: number analyzed (Participants) | 5
  1-<6 years | 6.47 (6.61)
  6-<12 years: number analyzed (Participants) | 5
  6-<12 years | 10.62 (9.06)
  Total | 8.54 (7.79)

11. Secondary Outcome: Spontaneous Annualized Bleeding Rate (SABR)
Description: The SABR was calculated in analogy to the TABR. The total number of spontaneous bleeding events (BEs) in the time period between the first dose of IMP and the study completion visit, divided by the duration (in years) between the first dose of IMP and the study completion visit.
  Surgery periods, and BEs occurring within these periods, will be excluded from the calculation of the SABR.
Time Frame: 6 months
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Spontaneous bleeding events per year
Arm/Group | Wilate
Number analyzed (Participants) | 10
Spontaneous bleeding events per year
  1-<6 years: number analyzed (Participants) | 5
  1-<6 years | 2.70 (2.93)
  6-<12 years: number analyzed (Participants) | 5
  6-<12 years | 1.20 (2.68)
  Total | 1.95 (2.76)

12. Secondary Outcome: Efficacy of Wilate in the Treatment of Breakthrough Bleeding Events (BEs)
Description: The proportion of BEs successfully treated with Wilate was assessed by the patient (together with the investigator in case of on-site treatment) in a patient diary. The treatment efficacy for all BEs was assessed using a pre-defined four-point scale: 'excellent', 'good', 'moderate', 'none'. 'Excellent' was defined as "Abrupt pain relief and/or unequivocal improvement in objective signs of bleeding within approximately 8 hours after a single injection" (best outcome); 'good 'was defined as "definite pain relief and/or improvement in signs of bleeding within approximately 8-12 hours after an injection, requiring up to 2 injections for complete resolution". All efficacy ratings assessed as either 'excellent' or 'good' were considered 'successfully treated'. 'Moderate' was defined as "probable or slight beneficial effect within approximately 12 hours after the first injection" and 'none' defined as "no improvement within 12 hours, or worsening of symptoms".
Time Frame: 6 months
Population: Analysis was performed in the per-protocol (PP) population. Of the patients in the PP population, only 8 patients had evaluable bleeding events. Five of these patients were aged 1-<6 years, and 3 aged 6-<12 years.
Measure: Count of Units; unit: Bleeding Events (BEs)
Units Other Than Participants: Bleeding Events (BEs)
Groups:
- 1-<6 Years: All patients in the PP population aged 1-<6 years.
- 6-<12 Years: All patients in the PP population aged 6-<12 years.
- Total: All patients in the PP population
Arm/Group | 1-<6 Years | 6-<12 Years | Total
Number analyzed (Participants) | 5 | 3 | 8
Number analyzed (Bleeding Events (BEs)) | 17 | 18 | 35
Bleeding Events (BEs)
  Excellent | 7 | 9 | 16
  Good | 9 | 8 | 17
  Moderate | 1 | 1 | 2
  None | 0 | 0 | 0

13. Secondary Outcome: Wilate Consumption Data: Average Dose of Wilate Per Week of Study
Description: The average consumption of Wilate per week of the study (IU/kg) for all patients receiving prophylaxis
Time Frame: 6 months
Population: The analysis was performed in the full analysis (FAS) population (total: n=10). The FAS comprised 5 patients were aged 1-<6 years and 5 were aged 6-<12 years.
Measure: Mean (Standard Deviation); unit: IU/kg per week
Groups:
- 1-<6 Years: All patients in the FAS population aged 1-<6 years.
- 6-<12 Years: All patients in the FAS population aged 6-<12 years.
- Total: Total patients in the FAS population
Arm/Group | 1-<6 Years | 6-<12 Years | Total
Number analyzed (Participants) | 5 | 5 | 10
IU/kg per week | 58.52 (14.85) | 68.08 (19.02) | 63.30 (16.86)

14. Secondary Outcome: Incremental in Vivo Recovery (IVR) of Wilate Over Time
Description: The rise in FVIII:C activity in IU/dl per unit dose administered in IU/kg was determined for all patients at baseline, 3 and 6 months, using the one-stage (OS) assay.
Time Frame: Baseline, and 3 and 6 months of treatment
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: kg/dL
Arm/Group | 1-<6 Years | 6-<12 Years | Total
Number analyzed (Participants) | 5 | 5 | 10
kg/dL
  Baseline | 1.65 (0.33) | 1.57 (0.53) | 1.61 (0.42)
  3 months | 1.55 (0.14) | 1.56 (0.57) | 1.56 (0.39)
  6 months | 1.63 (0.24) | 1.32 (0.45) | 1.48 (0.38)

15. Secondary Outcome: Association Between ABO Blood Type and the FVIII:C Half-life of Wilate (OS Assay)
Description: Analysis of variance (ANOVA) was used in an exploratory sense to assess a possible association between the ABO blood type and the FVIII:C half-life of Wilate. This was analysed by calculating the mean square in a one-stage (OS) assay.
Time Frame: 6 months
Population: The analysis was performed for the PK population which included all patients who underwent PK assessment during the study (total: n=10). The PK population comprised 5 patients aged 1-<6 years and 5 aged 6-<12 years.
Measure: Number; unit: Correlation coefficient
Arm/Group | Wilate
Number analyzed (Participants) | 10
Correlation coefficient
  1-<6 years: number analyzed (Participants) | 5
  1-<6 years | 0.185
  6-<12 years: number analyzed (Participants) | 5
  6-<12 years | 6.100
  Total | 0.922
Statistical Analysis 1: Comparison: Wilate; Test type: Other; p = 0.9593, ANOVA — P-Value for patients aged 1-<6 years (N=5)
Statistical Analysis 2: Comparison: Wilate; Test type: Other; p = 0.3752, ANOVA — P-Value for patients aged 6-<12 years (N=5)
Statistical Analysis 3: Comparison: Wilate; Test type: Other; p = 0.8273, ANOVA — P-Value for total PK population (N=10)

16. Secondary Outcome: Association Between VWF:Ag Concentration and the FVIII:C Half-life of Wilate
Description: Analysis of variance (ANOVA) was used in an exploratory sense to assess a possible association between VWF:Ag with the FVIII:C half-life of Wilate. This was analysed by calculating the mean square in a one-stage (OS) assay.
Time Frame: 6 months
Population: The analysis was performed for the PK population which included all patients who underwent PK assessment during the study (total: n=10).
Measure: Number; unit: Correlation coefficient
Arm/Group | Wilate
Number analyzed (Participants) | 10
Correlation coefficient
  1-<6 years: number analyzed (Participants) | 5
  1-<6 years | 0.121
  6-<12 years: number analyzed (Participants) | 5
  6-<12 years | 0.006
  Total | 0.003
Statistical Analysis 1: Comparison: Wilate; Test type: Other — P-Value for patients aged 1-<6 years (N=5); p = 0.8536, ANOVA
Statistical Analysis 2: Comparison: Wilate; Test type: Other; p = 0.9791, ANOVA — P-Value for patients aged 6-<12 years (N=5)
Statistical Analysis 3: Comparison: Wilate; Test type: Other; p = 0.9791, ANOVA — P-Value for total PK population (N=10)

17. Secondary Outcome: Safety and Tolerability of Wilate by Monitoring The Number of Adverse Events (AEs) Throughout the Study
Description: At each visit (whether scheduled or unscheduled) , AEs will be documented by the investigator throughout the study. In addition, the investigator will check the patient diaries for any documented event.
Time Frame: 6 months
Population: The safety (SAF) population included all patients who received at least one injection of Wilate during the study (n=10).
Measure: Number; unit: Adverse events
Groups:
- Wilate: The safety (SAF) population
Arm/Group | Wilate
Number analyzed (Participants) | 10
Adverse events | 6

18. Secondary Outcome: Immunogenicity of Wilate: Number of Participants With FVIII Inhibitor Activity at 6 Months
Description: FVIII inhibitor activity was determined at each study visit: screening, PK, Day 14 visit, Day 30 visit, 3 Months visit and 6 Months visit before injection.
Time Frame: 6 months
Population: The analysis was performed in the overall safety (SAF) population included all patients who received at least one injection of Wilate during the study (n=10). Of these, 5 patients 1-<6 years were analyzed, and 5 patients aged 6-<12 years were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Wilate
Number analyzed (Participants) | 10
Participants | 0
Statistical Analysis 1: Comparison: Wilate; Test type: Other; Pearson-Copper = 0, 95% CI 2-sided [0 to 30.85]

19. Secondary Outcome: Virus Safety Measured by the Number With Parvovirus B19 Seroconversions Between Baseline (BL) and End of Study
Description: Virus safety was evaluated by taking a plasma sample for parvovirus B19 antibody testing before the first injection of Wilate at the PK visit. All patients negative at screening were tested again at the Study Completion visit. The number of Parvovirus B19 seroconversions between BL and end of study was recorded
Time Frame: 6 months
Population: Analysis was performed in all patients who underwent full analysis (FAS population) (n=10).
Measure: Number; unit: Participants with seroconversions
Arm/Group | Wilate
Number analyzed (Participants) | 10
Participants with seroconversions | 1

ADVERSE EVENTS:
Time Frame: Between the screening visit and the follow up contact visit (30 days after the 6-month study completion visit)
Arm/Group | Wilate
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 1/10
Other Adverse Events (participants affected / at risk) | 3/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Wilate (N=10)
Cryptochidism (Congenital, familial and genetic disorders) | 1 (1) — One patient had a treatment emergent adverse event (TEAE) that was classified as serious because it required hospitalisation for surgery. The adverse event was judged as moderate and not related to Wilate.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Wilate (N=10)
Respiratory tract infection (Infections and infestations) | 1 (1)
Varicella (Infections and infestations) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Parvovirus B19 test positive (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-06-19): https://cdn.clinicaltrials.gov/large-docs/16/NCT03376516/Prot_002.pdf
  • Statistical Analysis Plan (2019-07-08): https://cdn.clinicaltrials.gov/large-docs/16/NCT03376516/SAP_003.pdf